CLINICAL TRIAL: NCT01120054
Title: Traumatic Brain Injury Among Homeless Veterans
Status: Completed | Type: Observational
Sponsor: VA Eastern Colorado Health Care System (U.S. Federal Agency)
Collaborators: US Department of Veterans Affairs (U.S. Federal Agency); Corporal Michael J. Crescenz VA Medical Center (U.S. Federal Agency); James A. Haley Veterans Administration Hospital (U.S. Federal Agency)
Responsible Party: Principal Investigator, Lisa Brenner, Director, VISN 19 MIRECC, VA Eastern Colorado Health Care System
Other Study IDs: 10-0170
Record Dates: First submitted 2010-05-06; First posted 2010-05-10 (Estimated); Last update posted 2019-01-31 (Actual); Status verified 2019-01

CONDITIONS: Traumatic Brain Injury; Homelessness
Keywords: Traumatic Brain Injury; Homelessness
MeSH Terms: conditions — Brain Injuries, Traumatic

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No

SUMMARY:
Objectives include: 1) establishing a psychometrically sound traumatic brain injury (TBI) screening measure for use among homeless veterans; 2) identifying the prevalence of those that screen positive for TBI among homeless veterans seeking VA services; and 3) comparing psychiatric and psychosocial outcomes between those with and without a history of TBI.

DETAILED DESCRIPTION:
Short-term Objectives include:

1. Establishing the criterion-related validity of the Traumatic Brain Injury-4 (TBI-4) questionnaire in the Veteran homeless population using the Ohio State University TBI-Identification Method (OSU TBI-ID) (Corrigan et al., 2007) as the gold standard for establishing traumatic brain injury (TBI) diagnosis.
2. Identifying the prevalence of those that screen positive for a lifetime history of TBI among homeless Veterans.
3. Comparing psychiatric outcomes (psychiatric hospitalizations, suicide attempts and deaths, and clinical contacts) and psychosocial outcomes between those with and without a lifetime history of TBI.

ELIGIBILITY:
Inclusion Criteria:

* At least 18 years of age, seeking homeless services at one of the VA Homeless Services Programs.

Exclusion Criteria:

* Failure to provide informed consent, not older than 89 years of age.

Ages: 18 Years to 89 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Homeless Veterans
Sampling Method: Non-Probability Sample
Enrollment: 2000 (Estimated)
Dates: Start 2010-05 (Actual); Primary Completion 2018-12 (Actual); Study Completion 2018-12 (Actual)

PRIMARY OUTCOMES:
OSU TBI-ID | One Time
  History of TBI

CONTACTS AND LOCATIONS:
Overall Officials: Lisa A. Brenner, Ph. D., Principal Investigator — VISN 19 MIRECC
Locations (3):
- United States (3):
  - Department of Veterans Affairs, Eastern Colorado Health Care System, Denver, Colorado
  - Tampa VAMC, Tampa, Florida
  - Philadelphia VAMC, Philadelphia, Pennsylvania

REFERENCES:
- See also: MIRECC Web Site — https://www.mirecc.va.gov/visn19/trm/